CLINICAL TRIAL: NCT02101047
Title: Correlation and Effects on Cardiac Output With Intermittent Phenylephrine Administration of 50 mcg Versus 100 mcg or 100mcg/Min Prophylactic Infusion for Treatment of Hypotension in Parturients After Receiving Spinal Anesthesia for Cesarean Delivery
Brief Title: Phenylephrine Dose and Mode of Administration for Spinal Anesthesia Induced Hypotension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of eligible participant
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 26872
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-02

CONDITIONS: Complications; Cesarean Section; Spinal Anesthetics Causing Adverse Effects in Therapeutic Use
Keywords: cesarean section; hypotension; phenylephrine
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- phenylephrine 50mcg bolus (Experimental): Phenylephrine 50 mcg bolus dosing with continuous placebo infusion
  Interventions: Drug: Phenylephrine
- Phenylephrine 100 mcg bolus (Experimental): Phenylephrine 100 mcg bolus dosing wtih continuous placebo infusion.
  Interventions: Drug: Phenylephrine
- Phenylephrine continuous infusion 100mcg/min (Experimental): Continuous phenylephrine infusion of 100 mcg/min with placebo bolus dosing.
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Phenylephrine

SUMMARY:
Three different regimens of phenylephrine are being evaluated to see if one is superior over the other in the maintenance of cardiac output while keeping normotension and/or treating hypotension experienced when receiving spinal anesthesia for cesarean delivery.

DETAILED DESCRIPTION:
Phenylephrine will be administered in one of 3 regimens: Intermittent bolus of 50 mcg, Intermittent bolus of 100 mcg, or continuous infusion of 100 mcg/min. The infusion will contain either phenylephrine or normal saline (placebo). Subjects who are randomized to receive a bolus dose will receive placebo in the infusion. Subjects who are randomized to receive the phenylephrine infusion will have normal saline (placebo) in the bolus syringe. Baseline blood pressures will be obtained prior to surgery and then maintained using these drugs. Blood pressure and heart rate will be monitored as usual standard of care. Continuous cardiac output and hemodynamic monitoring will be obtained using CNAP (Tm) or similar (equivalent) monitoring device. Blood pressure will be maintained at 90-120% of baseline utilizing infusion and/or bolus with the 3 regimens.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for cesarean delivery age >/=18 years of age >/= 37 weeks EGA ASA status I-III

Exclusion Criteria:

* allergy to medications used in the study non-English speaking

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Magnitude of cardiac output changes | 0-90 minutes
  Magnitude of cardiac output reduction for the duration from preoperative baseline from time of spinal anesthesia to delivery of fetus and placenta.

SECONDARY OUTCOMES:
provider intervention | 0-90 minutes
  number of provider intervention to treat abnormal hemodynamics
vasopressor requirement | 0-90 minutes
  total amount of vasopressor or equivalent required
Emetic symptoms | 0-90 minutes
  emetic symptoms - magnitude and/or incidence
hypertension | 0-90 minutes
  incidence and magnitude
hypotension | 0-90 minutes
  incidence and magnitude
bradycardia | 0-90 minutes
  incidence and magnitude
Anesthetic time | up to 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pan, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Novant Health Forsyth Medical Center, Winston-Salem, North Carolina, United States